CLINICAL TRIAL: NCT01279707
Title: Phase I/II Study Combining Humanised Anti-CD20 (Veltuzumab), Anti-CD22 (Epratuzumab) and Both Monoclonal Antibodies With Intensive Chemotherapy in Adults With Recurrent or Refractory B-precursor Acute Lymphoblastic Leukaemia (ALL)
Brief Title: Monoclonal Antibodies in Recurrent or Refractory B Cell Acute Lymphoblastic Leukaemia (ALL) (MARALL)
Acronym: MARALL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6125
Record Dates: First submitted 2010-04-12; First posted 2011-01-19 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Recurrent or Refractory B Cell Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma | interventions — veltuzumab; epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: Veltuzumab and chemotherapy (Experimental): Veltuzumab and modified UKALL XII chemotherapy
  Interventions: Biological: humanised monoclonal antibody, veltuzumab
- B: epratuzumab and chemotherapy (Experimental): epratuzumab and modified UKALL XII chemotherapy
  Interventions: Biological: humanised monoclonal antibody epratuzumab
- C: veltuzumab and epratuzumab and chemotherapy (Experimental): Veltuzumab and Epratuzumab and modified UKALL XII chemotherapy
  Interventions: Biological: humanised monoclonal antibodies veltuzumab and epratuzumab

INTERVENTIONS:
Biological: humanised monoclonal antibody, veltuzumab — Veltuzumab with modified UKALL XII induction chemotherapy. Veltuzumab will be administered at 200 mg/m2 IV on Day 8 and subsequently, (if tolerated on Day 8), over 1 hour on Days 15, 22, 29.
  Arms: A: Veltuzumab and chemotherapy
Biological: humanised monoclonal antibody epratuzumab — Epratuzumab with modified UKALL XII induction chemotherapy. Epratuzumab will be administered at 360 mg/m2 IV over 1 hour on Days 8, 15, 22 and 29.
  Arms: B: epratuzumab and chemotherapy
Biological: humanised monoclonal antibodies veltuzumab and epratuzumab — Epratuzumab + Veltuzumab with modified UKALL XII induction chemotherapy. Epratuzumab will be administered at 360 mg/m2 IV over 1 hour on Days 8, 15, 22 and 29. Veltuzumab will be administered at 200 mg/m2 IV over 2 hours on Day 8 and over 1 hour on Days 15, 22 and 29. Veltuzumab will be infused 1 hour after the infusion of epratuzumab.
  Arms: C: veltuzumab and epratuzumab and chemotherapy

SUMMARY:
The treatment of adult B-cell acute lymphoblastic leukaemia (ALL) has progressed considerably in the past 3 decades, particularly due to intensification of chemotherapies, improved supportive care and the incorporation of stem cell transplantation. However, the maximum tolerability of standard chemotherapeutics has been reached in ALL. Using conventional chemotherapy, 80-85% of adults with ALL will achieve a complete remission (CR). Unfortunately treatment at relapse is generally unsuccessful and rarely results, in long-term survival (7% survival at 5 years). Therefore, the investigators are exploring novel treatment strategies through the use of monoclonal antibodies (MoAbs) directed at surface antigens on leukaemic blasts. Using MoAbs directed against surface proteins on B cells has had excellent results in other B-cell diseases such as low and high grade non-Hodgkin lymphomas, without additional toxicity. There has also been limited evidence from small studies and case reports of the efficacy of MoAbs in ALL.

This is a Phase I/II study to determine the safety and tolerability of the combination of veltuzumab and epratuzumab with intensive chemotherapy in patients with relapsed B-cell ALL. A maximum of 51 patients will be treated with a combination of UKALL XII induction chemotherapy and the monoclonal antibodies veltuzumab and epratuzumab. Veltuzumab and epratuzumab are humanised monoclonal antibodies that target CD20 and CD22 surface proteins, respectively. Both of these proteins are expressed on ALL tumour B cells.

One group of patients will receive modified UKALL XII chemotherapy + veltuzumab; a second, modified UKALL XII chemotherapy + epratuzumab and if limited toxicity is found in these first 2 groups, a third group will receive, modified UKALL XII chemotherapy + both veltuzumab and epratuzumab. Patients will be assessed for safety, tolerability and disease response. Safety and tolerability will be measured by the number of Dose Limiting Toxicities (DLTs) in each group. Disease response will be measured by the microscopic appearance of patient bone marrow samples at day 29, and by molecular tests for tumour cells in bone marrow.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 years or over
2. Confirmed diagnosis of recurrent or refractory B-precursor ALL [according to the WHO classification].
3. Greater than 5% blasts in the bone marrow
4. WHO/ECOG performance status of 0-2 and well enough to receive intensive combination chemotherapy.
5. Negative pregnancy test in women of childbearing potential. Women will not be considered of child bearing potential if they have undergone surgical removal of the uterus or are post menopausal and have been amenorrhoeic for at least 24 months.
6. Patients must have adequate organ function:

   * Renal function - serum creatinine <2.5 x ULN or eGFR>50ml/min (measured EDTA or estimated creatinine clearance e.g Cockcroft & Gault)
   * Liver function (bilirubin/ALT <2.5 x ULN)
7. Patients must be able to comply with the study schedule.

Exclusion Criteria:

1. Patients should not have received chemotherapy for current episode of relapsed ALL (except corticosteroids for a maximum of 10 days, before joining the study).
2. Patients with co-morbidities: e.g. uncontrolled hypertension and or poorly controlled diabetes which in the PI's opinion makes them unsuitable for the study.
3. Patients with severe psychiatric disorders which in the PI's opinion makes them unsuitable for trial participation.
4. Females of childbearing potential and all males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) for the duration of the study and for up to 3 months after the last dose of study medication. Note: Subjects are not considered of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
5. Females of childbearing potential must have a negative pregnancy test within 7 days prior to starting the study.
6. Females must not be breastfeeding.
7. Patients may not receive any other investigational agent during the study.
8. Patients should not have received any antibody therapy within 3 months of joining this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The total number of dose limiting toxicity events (DLTs) to measure safety and tolerability | Day 29
  The primary objective is to assess the safety and tolerability of the combination of veltuzumab and/or epratuzumab with intensive chemotherapy for recurrent or refractory adult B-precursor ALL.

SECONDARY OUTCOMES:
Morphological and molecular remission in bone marrow | Day 29
  Achievement of morphological complete remission on Day 29 bone marrow
  Efficacy of treatment to achieve MRD negativity, and investigate a possible association between the intensity of CD20 and CD22 antigen expression and treatment activity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, Doctor, Principal Investigator — Barts and The London NHS Trust
Locations (10):
- United Kingdom (10):
  - University Hospitals Birmingham NHS Foundation, Birmingham
  - University of Bristol Foundation Trust, Bristol
  - University Hospital of Wales, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Barts and the London NHS Trust, London
  - Royal Free Hampstead NHS Trust, London
  - Newcastle University, Newcastle
  - Nottingham City Hospital, Nottingham
  - Plymouth Hospitals NHS Trust, Plymouth